CLINICAL TRIAL: NCT06853470
Title: Safety and Efficacy of the SynFlow 3.0 Percutaneous Transvalvular Ventricular Assist System in Patients Undergoing High-Risk PCI: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Trial (PERSIST Ⅲ Study)
Brief Title: Prospective Evaluation for Receiving SynFlow 3.0 Interventional Circulatory Support in High-risk PCI: A Randomized Controlled Trial
Acronym: PERSIST Ⅲ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ForQaly Medical (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRPR002
Record Dates: First submitted 2025-02-19; First posted 2025-03-03 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: High Risk PCI; Coronary Arterial Disease (CAD)
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SynFlow3.0 (Experimental): The patients will undergo PCI and use SynFlow3.0 as hemodynamic supoort during the PCI
  Interventions: Device: SynFlow 3.0 circulatory support; Procedure: percutaneous coronary intervention
- V-A ECMO (Active Comparator): The patient will receive PCI and use V-A ECMO as hemodynamic support during the PCI
  Interventions: Device: VA-ECMO circulatory support; Procedure: percutaneous coronary intervention

INTERVENTIONS:
Device: VA-ECMO circulatory support — Venoarterial extracorporeal membrane oxygenation (VA-ECMO) is a percutaneous mechanical circulatory support device that can provide short-term hemodynamic support during high-risk PCI.
  Arms: V-A ECMO
Device: SynFlow 3.0 circulatory support — The SynFlow 3.0 is a novel percutaneous left ventricular-assist device that can provide temporary hemodynamic support during high-risk procedure.
  Arms: SynFlow3.0
Procedure: percutaneous coronary intervention — The percutaneous coronary intervention is a percutaneous endovascular intervention technique that can restore coronary blood flow by various intervention methods such as angioplasty and stent implantation.

SUMMARY:
This study is conducted to compare the effectiveness of a new percutaneous mechanical circulatory support device called SynFlow 3.0 with VA-ECMO in high-risk percutaneous coronary intervetnion(PCI) patients. The objective of this study is to see if SynFlow 3.0 can provide similar or better support during high-risk PCI compared to VA-ECMO.

Specifically, the following questions is to be answered in this study:

Can SynFlow 3.0 provide sufficient hemodynamic support for patients during high-risk PCI and the effect be similar to VA-ECMO? Does SynFlow 3.0 offer other clinical benefits compared to VA-ECMO? By answering these questions, it will be determined if SynFlow 3.0 can be a viable alternative to VA-ECMO for patients undergoing high-risk PCI.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, randomized controlled trial under the Good Clinical Principles(GCP) carried out in more than 15 research centers over China. Patients with 3-vessel disease, unprotected left main coronary artery disease or last patent conduit and severly depressed left ventricular function (LVEF≤35%) will be enrolled and undergo non-emergent PCI, and be randomized 1:1 to receive either the SynFlow 3.0 or VA-ECMO support during the PCI. The primary endpoint is the incidence of 30-day major adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The investigator assesses that the subject requires coronary revascularization, but CABG is considered as high-risk or the subject refuses CABG. The investigator considers the subject may benefit from PCI.
2. Left ventricular ejection fraction (LVEF) ≤ 35%.
3. Coronary angiography (CAG) or coronary computed tomography angiography (CTA) shows any of the following conditions:

   1. last patent conduit (occluded vessel diameter ≥ 2.5 mm).
   2. unprotected left main (LM) coronary artery disease.
   3. Three-vessel disease (stenosis ≥ 70%). *Three-vessel disease is defined as at least one significant stenosis (≥ 70%) lesion in all three major epicardial coronary artery territories: left anterior descending artery (LAD) and/or its branches, left circumflex artery (LCX) and/or its branches, and right coronary artery (RCA) and/or its branches. In the case of left coronary artery dominance, a lesion in the LAD and the proximal LCX qualified as three-vessel disease.
4. The subject is able to understand the purpose of the trial and sign the informed consent form, and is likely to be compliant to and willing to receive the clinical follow up after discharge.

Exclusion Criteria:

1. STEMI within 24 hours.
2. Cardiac arrest within 24 hours.
3. Cardiogenic shock (CS) or acute decompensation of chronic heart failure (Cardiogenic shock is defined as systemic hypotension [systolic blood pressure <90 mmHg or requiring inotropes/vasopressors to maintain systolic blood pressure >90 mmHg] and any of the followings: ongoing need for inotropes/vasopressors before entering the catheterization lab, any clinical evidence of end-organ hypoperfusion, or use of IABP or other circulatory support devices).
4. History of stroke or TIA within one month prior to the procedure.
5. Contraindications to or inability to place pVAD and ECMO (including but not limited to: left ventricular thrombus, presence of a mechanical aortic valve or cardiac contractile device, moderate to severe aortic stenosis, moderate to severe aortic regurgitation, stents in peripheral access or severe peripheral vascular disease such as tortuosity and dissection which impedes device placement, aortic dissection, aortic aneurysm, or severe abnormalities of ascending aorta or aortic arch , hematological diseases causing fragility of blood cells or hemolysis , hypertrophic obstructive cardiomyopathy).
6. Presence or suspicion of active systemic infection.
7. Known contraindications to heparin (including heparin-induced thrombocytopenia), contrast agents, or study-required medications (e.g., aspirin, clopidogrel).
8. Uncorrectable coagulopathy prior to the procedure, including platelet count ≤75×10^9^/L or INR ≥2.0.
9. Liver dysfunction: liver enzymes and bilirubin of more than 3 times the upper limit of the normal value.
10. Renal dysfunction: undergoing dialysis or serum creatinine ≥4 mg/dL (353.6 µmol/L).
11. Severe right heart failure or severe tricuspid regurgitation.
12. Pregnant or lactating women, or women planning pregnancy during the trial.
13. Participation in another drug or medical device clinical trial without reaching the primary endpoint.
14. Other conditions deemed by the investigator as unsuitable for participation in this trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Adverse Events (MAE) | Up to 30 days

SECONDARY OUTCOMES:
Incidence of MAE | Up to 90 days
Incidence of major adverse cardiac and cerebral events (MACCE) | Up to 30 days, up to 90days
the change of left ventricular ejection fraction (LVEF) compared to baseline | before discharge, at 30±7 days, at 90±14 days
the change of New York Heart Association (NYHA) class compared to baseline | before discharge, at 30±7 days, at 90±14 days
Total length of hospital stay | Up to 30 days
ICU/CCU length of stay | Up to 30 days
Incidence of adverse events | Up to 90 days
Incidence of serious adverse events | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Phd, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Dan Song, Phd, Principal Investigator — Wuhan Asia Heart Hospital; Bo Luan, Phd, Principal Investigator — Liaoning Provincial People's Hospital; Chuanyu Gao, Phd, Principal Investigator — Fuwai Huazhong Cardiovascular Hospital; Cheng Zhang, Phd, Principal Investigator — Qilu Hospital of Shandong University; Jingping Wang, Phd, Principal Investigator — Shanxi Cardiovascular Hospital; Zuyi Yuan, Phd, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yining Yang, Phd, Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; Yan Wang, Principal Investigator — Xiamen Cardiovascular Hospital; Yan Li, Phd, Principal Investigator — The Second Affiliated Hospital of Air Force Medical University; Yansong Guo, Phd, Principal Investigator — Fujian Provincial Hospital; Ming Bai, Phd, Principal Investigator — LanZhou University; Renqiang Yang, Phd, Principal Investigator — Second Affiliated Hospital of Nanchang University; Jiancheng Xiu, Phd, Principal Investigator — Nanfang Hospital, Southern Medical University; Jianhong Tao, Phd, Principal Investigator — Sichuan Academy of Medical Sciences; Min Dai, Phd, Principal Investigator — Mianyang Central Hospital; Lin Zhao, Phd, Principal Investigator — Beijing Chao Yang Hospital; Yundai Chen, Phd, Study Chair — First Medical Center of the General Hospital of the People's Liberation Army; Junbo Ge, Phd, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China